CLINICAL TRIAL: NCT05823311
Title: A Randomized, Double-blind, Multicenter Study of Lenvatinib, Temalizumab Combined with Gemcitabine and Cisplatin (GPLET) in the Treatment of Advanced Cholangiocarcinoma
Brief Title: Lenvatinib, Tislelizumab Combined with Gemcitabine and Cisplatin (GPLET) in the Treatment of Advanced Cholangiocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Tumor Hospital of Xinjiang Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0175
Record Dates: First submitted 2023-03-12; First posted 2023-04-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cholangiocarcinoma
Keywords: Lenvatinib; Tislelizumab; Gemcitabine and Cisplatin
MeSH Terms: interventions — lenvatinib; tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GPLET (Lenvatinib, Tislelizumab Plus Gemcitabine and Cisplatin) (Experimental): Intravenous injection: gemcitabine and cisplatin (CG)+ tislelizumab； Oral administration: lenvatinib.
  Interventions: Drug: Lenvatinib, tislelizumab, gemcitabine and cisplatin
- CG (Gemcitabine and Cisplatin) (Placebo Comparator): Intravenous injection: gemcitabine and cisplatin (CG)+placebo； Oral administration: placebo.
  Interventions: Drug: Gemcitabine and cisplatin

INTERVENTIONS:
Drug: Lenvatinib, tislelizumab, gemcitabine and cisplatin — Intravenous injection: gemcitabine and cisplatin (CG) + tislelizumab； Oral administration: lenvatinib.
  Arms: GPLET (Lenvatinib, Tislelizumab Plus Gemcitabine and Cisplatin)
Drug: Gemcitabine and cisplatin — Intravenous injection: gemcitabine and cisplatin (CG) + placebo； Oral administration: placebo.
  Arms: CG (Gemcitabine and Cisplatin)

SUMMARY:
Cholangiocarcinoma (CCA) is a heterogeneous group of cancers arising from the epithelial cells of bile ducts. Because of highly aggressive malignancy, most of the patients are diagnosed at an advanced stage and lose the chance to undergo surgery.

As more effective and novel chemotherapy, targeted therapies, and immunotherapy become available, multiple treatments can be chosen for the patients with advanced CCA. Cytotoxic cell death during tumor chemotherapy triggers antigen release and induces strong anti-tumor effects of T cells. Tyrosine kinase inhibitors (TKI) can reduce the expression of PD-L1 and inhibit Treg cell infiltration, and together with immune checkpoint inhibitors, they can relieve tumor immunosuppressive microenvironment.

Therefore, the study aims to investigate the safety and efficacy of Lenvatinib, Tislelizumab combined with Gemcitabine plus Cisplatin (GPLET) in the treatment of advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, unresectable advanced or metastatic cholangiocarcinoma patients.
* Expected survival period > 12 weeks.
* The World Health Organization (WHO) / ECOG physical status (PS) was 0 or 1.
* There was at least one target lesion that matched the RECIST 1.1 criteria at baseline.
* Not previously received immunotherapy, including but not limited to CTLA 4, PD-L1 or/and PD-1 inhibitors.
* Adequate organ and bone marrow function, defined as follows: Hemoglobin (Hb)≥9.0g/dL; Neutrophils (ANC) ≥ 1.5* 10^9/L; Platelet (Pt) ≥ 50*10^9/L; ALT≤2.5×ULN（Normal upper limit); AST≤2.5×ULN.
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Active or previously documented autoimmune disease or inflammatory disease.
* Uncontrolled complications.
* History of other primary malignancies.
* Active infection.
* Women who are pregnant or breastfeeding.
* Patients with severe allergic history or specific constitution.
* Researchers consider it inappropriate to participate in the test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | At the end of 4 treatment cycles(each cycle is 21 days)
  The proportion of patients with at least one complete response (CR) or partial response (PR) (%)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression, assessed up to 60 months
  The time between the date of randomization and the date of radiographic progression
Overall survival time (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  The time between the date of randomization and death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China